CLINICAL TRIAL: NCT04101877
Title: The Sahlgrenska Anti-VEGF (SAHLVE) Study - a Prospective Randomized Double-blind Comparison of Bevacizumab and Aflibercept in Patients With Neovascular Age-related Macular Degeneration
Brief Title: The Sahlgrenska Anti-VEGF Study
Acronym: SAHLVE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAHLVE; 2018-004438-14 (EudraCT Number)
Record Dates: First submitted 2019-09-13; First posted 2019-09-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — Bevacizumab; aflibercept

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, randomized, double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avastin (Experimental): bevacizumab 25 mg/ml, intravitreal administration, 0.05 ml (1.25 mg)
  Interventions: Drug: Bevacizumab Injection
- Eylea (Active Comparator): aflibercept 40 mg/ml, intravitreal administration, 0.05 ml (2 mg)
  Interventions: Drug: Aflibercept Injection

INTERVENTIONS:
Drug: Bevacizumab Injection — 25 mg/ml
  Other Names: Avastin
  Arms: Avastin
Drug: Aflibercept Injection — 40 mg/ml
  Other Names: Eylea
  Arms: Eylea

SUMMARY:
The study investigates whether patients treated for neovascular (wet) age-related macular degeneration (AMD), with intravitreal injection with bevacizumab (Avastin) after two years need more injections with retained therapy response compared to patients being treated with intravitreal injection with aflibercept (Eylea).

The study also aims to evaluate if there is a difference in best-corrected visual acuity, macular thickness, recurrence interval, durability, cost efficiency, as well as vision-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent.

≥50 years, regardless of gender.

Diagnosed with the neovascular (wet) form of age-related macular degeneration through diagnosed neovascular vascular membranes with OCT-A and, if necessary, also FA / ICG, according to clinical routine.

Distance visual acuity ≥34 (ETDRS) on the current study eye.

Exclusion Criteria:

Other eye disease in the current study eye that affects visual acuity or the possibility of examining fundus, according to the investigator's assessment.

Previously received treatment for the neovascular (wet) form of age-related macular degeneration.

Diagnosed with diabetes (all types).

Degenerative state of the macula that prevents vision improvement such as central areolar atrophy or other pronounced dry AMD or fibrosis, in the current study eye.

Other choroidal neovascularization (CNV) of the type PCV or due to grave myopia i.e. ≥ 6.0 diopters (D) or secondary to other retinal disease, in the current study eye.

Unregulated intraocular pressure (IOP) > 30 mmHg despite pharmacological treatment in the current study eye.

Have had a stroke or heart attack ≤6 months ago.

Inability to access information (e.g. due to dementia) or inability to conduct examinations (e.g. ETDRS examination), according to the investigator's assessment.

Inability to receive oral and written information in Swedish (in need of an interpreter).

Included in another intervention study.

Fertile woman i.e. a woman who has had menstruation for the past 12 months or has not undergone permanent sterilization (hysterectomy, bilateral salpingectomy or bilateral oophorectomy).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of injections | Two years
  Number of intravitreal injections

SECONDARY OUTCOMES:
Best-corrected visual acuity (BCVA), distance | Two years
  ETDRS
Best-corrected visual acuity (BCVA), near | Two years
  LIX
Macular thickness (Central Retinal Thickness; CRT) | Two years
  μm
Intraocular pressure (IOP) | Two years
  mmHg
Recurrence interval | Two years
  Maximum number of weeks from last injection to relapse, at first and last relapse.
Durability | Two years
  Longest inactive interval detected (number of weeks).
Cost efficiency | Two years
  Quality-adjusted life years (QALY), cost-per-QALY is measured with the EuroQol-5 Dimension (EQ-5D) questionnaire.
  EQ-5D consists of five subscales: mobility, self-care, usual activities, discomfort/pain and anxiety/depression. The subscales measure different aspects of health and well-being where the subject is asked to rank each subscale from 1 (no problems) to 3 (major problems). These answers are converted to a score between 0 (=death) to 1 (=full health). The subscales are converted to a weighted mean which ranges from 0 (death) to 1 (full health). Negative values may exists for conditions worse than death. The weighting differs between geographic areas; for Sweden, the UK weighting scale is used.
Vision-related quality of life | Two years
  National Eye Institute Visual Functioning Questionnaire -25 (NEI VFQ-25) questionnaire is based on 25 questions (items) where the subject is asked questions on visual function, daily activities and social consequences of visual function. The questions have answers on a 5- or 6-grade scale which are converted to a scale from 0 (no function/worst consequence) to 100 (no problems). The 25 items are clustered into 12 subscales. Items within each subscale are averaged to create the subscale scores according to the NEI VFQ-25 scoring algorithm. In addition, a composite score for all 12 subscales are created as an average of these. Minimum score is 0 and maximum score is 100 for each item, subscale and the composite score.
Cost-benefit | Two years
  The incremental cost-effectiveness ratio (ICER) is a statistic used in cost-effectiveness analysis to summarise the cost-effectiveness of a health care intervention. It represents the average incremental cost associated with 1 additional unit of the measure of effect and is given in Euro.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Zetterberg, MD, PhD, Principal Investigator — Vastra Gotaland Region
Locations (1):
- Vastra Gotaland Region, Sahlgrenska University Hospital, Department of Ophthalmology, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, however, the results (group-level) will be available within one year of study completion.